CLINICAL TRIAL: NCT04852211
Title: Asia-Pacific Multi-Centre Randomized Trial of Laparoscopic Versus Open Major Hepatectomy for Hepatocellular Carcinoma (AP-LAPO Trial)
Brief Title: Laparoscopic Versus Open Major Hepatectomy for HCC Hepatectomy for Hepatocellular Carcinoma
Acronym: AP-LAPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medicine Research Fund (Unknown)
Responsible Party: Principal Investigator, Kelvin K.C. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002kkcng/surg/cuhk
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Laparoscopic surgery; Open Surgery; Major hepatectomy; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Patients with hepatocellular carcinoma which undergone major hepatectomy will be randomized to either laparoscopic or open surgery group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open major hepatectomy (Active Comparator): Resection of the tumor together with 3 or more liver segments using open standard techniques of hepatectomy
  Interventions: Procedure: Open or laparoscopic surgery
- Laparoscopic major hepatectomy (Active Comparator): Resection of the tumor together with 3 or more liver segments using minimally invasive techniques of hepatectomy
  Interventions: Procedure: Open or laparoscopic surgery

INTERVENTIONS:
Procedure: Open or laparoscopic surgery — Patients, with their consent, will be recruited to participate by investigators after considering the inclusion and exclusion criteria. Treatment allocation to the eligible patients will follow a randomization schedule. A total of 212 subjects will be randomized 1:1 to one of the two treatment arms:
  1. Laparoscopic group: LMH
  2. Open group: OMH

SUMMARY:
Background: Hepatocellular carcinoma (HCC) is the sixth most common malignancy in the world. Major hepatectomy (resection of > 3 liver segments) is needed if tumor is close to major blood vessels within liver. Despite low mortality, open major hepatectomy (OMH) is associated with high tumor recurrence rate, and short survival. Immunosuppression due to surgical stress and blood transfusion, and dissemination of tumor cells because of tumor manipulation all contribute to tumor recurrence.

Laparoscopic major hepatectomy (LMH) is a newly developed minimally invasive technique for HCC. Apart from less wound problems and shorter recovery time than open surgery, LMH may have potential oncological benefits of prolonging survival. These could be related to the reduced intraoperative blood loss, less immunosuppression due to surgical stress, and less tumor manipulation. Hence, LMH could be a better treatment option than OMH for HCC.

Objectives:

1. To compare the long-term oncological outcome between laparoscopic and open major hepatectomy for patients with hepatocellular carcinoma
2. To achieve the comparison under the study design of multi-center randomized trial involving 5 high-volume centers in Asia-Pacific region
3. Primary outcome is 2-year recurrence-free survival.
4. Secondary outcome as intraoperative blood loss, blood transfusion, 30-day and hospital mortality, postoperative morbidities according Clavien-Dindo classification, hospital stay, quality of life, overall and recurrence-free survival rates up to 5 years after surgery
5. To compare the perioperative changes in stress-related cytokines, which help to clarify the stress response and immunosuppression and their correlations with overall and recurrence-free survival rates

Hypothesis: Laparoscopic major hepatectomy is associated with less surgical stress, less immunosuppression and thus less tumor recurrence and better survival than open major hepatectomy.

Study design: This is an open-labelled prospective randomized trial involving 106 patients in each treatment arm (Total number of patients recruited: 212). The study will involve 5 surgery centers in Asia-Pacific region (2 centers in Hong Kong, 3 centers in Mainland China Foshan, Shanghai and Sichuan).

Subjects: Patients with HCC undergone major hepatectomy. Recruitment centres involved:

1. Department of Surgery, The Chinese University of Hong Kong
2. Department of Surgery, Kwong Wah Hospital, Hong Kong
3. Department of Surgery, West China Medical School of Sichuan University
4. Department of Biliary Surgery, Eastern Hepatobiliary Surgery Hospital & Institute, Second Military Medical University
5. Department of Surgery, The First People's Hospital of Foshan

Intervention: Consented patient will be randomized 1:1 to one of the two treatment arms:

1. Laparoscopic group: LMH
2. Open group: OMH The randomization schedule will be generated by the Clinical Trials Centre (CTC) of principle investigator's center, prior to the start of the study.

Main outcome measure: The primary objective is to test the hypothesis that LMH is associated with less surgical stress, less immunosuppression and thus less tumor recurrence and better survival than OMH. The primary outcome measure is 2-year recurrence-free survival.

Data analysis: Statistical plan and data monitoring Statistical analysis will be performed using SPSS version 11.0 (SPSS Inc., Chicago, Ill). The 2-year recurrence-free survival (primary outcome) will be evaluated by Kaplan-Meier method and compared by the log-rank test between studied groups.

Expected results: The result of this study provides level 1 evidence on the best treatment option for HCC, which needs major hepatectomy. Such information will influence the evidence-based policy in professional practice in the management algorithm for HCC. Since postoperative complications and tumor recurrence are substantial after OMH, potential benefits of LMH tested in this study will help to alleviate these problems.

DETAILED DESCRIPTION:
Background: Hepatocellular carcinoma (HCC) is the sixth most common malignancy in the world.The practice of screening by ultrasonography and serum alpha-fetoprotein concentration in cirrhotic patients and hepatitis B carriers has led to an increasing incidence of HCC.

Hepatectomy, local ablation and liver transplantation are regarded as the mainstay of curative treatment for HCC according to international guidelines by EASL, AASLD and ESMO.The shortage of liver grafts has limited the application of liver transplantation. Hepatectomy is thus widely accepted as the treatment option of choice for patients with HCC and non cirrhotic liver.

Major hepatectomy (resection of > 3 Couinaud's segments) is always needed when HCC is large or is close to major blood vessels within liver. With the advancements in techniques of hepatectomy and perioperative patient care, the operative mortality of open major hepatectomy (OMH) has reduced to < 5% in recent years. Nonetheless, OMH for HCC is still associated with major problems as follows:

1. It is associated with significant morbidities. The morbidity rate after OMH remains high (30% - 40%) even in high-volume centres. Wound infection and bronchopneumonia are among the most common complications after hepatic resection. Long incision and vigorous retraction of the rib cage are required to achieve adequate exposure of the liver tumor during hepatic resection. As a result, sepsis due to chest complications and wound problems are frequently encountered. Furthermore, division of the porto-systemic collaterals in the anterior abdominal wall contributes to postoperative ascites, which is another common complication.
2. It is associated with a high tumor recurrence rate, even when performed with a curative intent. The 3-year recurrence rate has been reported to be more than 50%. Most recurrences occur in the liver remnant, in the forms of intrahepatic metastasis or multicentric tumor recurrence. Risk factors related to recurrence include unfavorable tumor factors such as microscopic venous or capsular invasion. Hence, tumor cell dissemination could be the main mechanism of recurrence. In this context, manipulation of the tumor during OMH leading to tumor cell dissemination can potentially contribute to high tumor recurrence rate. Furthermore, it has been suggested that postoperative immunosuppression induced by surgical stress may induce tumor growth in the liver remnant.

Laparoscopy has a well-defined role in the staging and diagnosis of hepatobiliary malignancies. However, laparoscopic hepatectomy has not yet been widely practiced, because of the technical difficulties in liver resection, difficulty in the control of hemorrhage during liver transection and retraction of the liver for optimum exposure. With the advanced laparoscopic techniques, much enthusiasm has been developed in laparoscopic major hepatectomy (LMH). Recent series have proven the feasibility and safety of LMH for HCC. The selection criteria of the reported series included tumor size up to 10cm and single or multiple tumors confined to one liver lobe. The overall conversion rates was around 10%. There was no hospital mortality and the morbidity rate was about 10%. Apart from the documented advantages of laparoscopic surgery (less wound and chest complications, and shorter hospital stay), theoretically, LMH carries oncological advantages over OMH. LMH may result in less surgical stress and immunosuppression due to less intraoperative blood loss than OMH. Moreover, using laparoscopic instruments, it involves minimal manipulation of the tumor and less cancer cells dissemination during surgery. Potentially, postoperative tumor recurrence could be reduced and hence patient survival could be prolonged.

To date, only retrospective studies using propensity score matching to compare LMH with OMH were reported. In these study, the studied patient number was small (< 40) in each matched treatment arm and the reported 2-year overall (86% - 88% vs. 85% - 100%) and recurrence-free survival (72% - 83% vs. 81% - 85%) rates were comparable between OMH and LMH. Nevertheless, there is a trend that LMH is associated with better overall and recurrence-free survival than OMH. It is likely that these studies were underpowered (Type II error) to show the potential oncological benefits of LMH over OMH. Because of these limited data on LMH, according to EASL, AASLD and ESMO guidelines, its role for HCC is still not yet defined. In the sphere of laparoscopic hepatectomy, according to the European Guideline Meeting for Laparoscopic Liver Surgery (Southampton consensus), there was only limited data on short-term outcome but no data on long-term outcome of LMH. With these reasons, there is an urge for a prospective study aiming to define the role of LMH for HCC with respect to its potential oncological benefits.

In the principle investigator's institution (the Department of Surgery, The Chinese University of Hong Kong), preliminary data using propensity score matching analysis on patients with HCC (median size = 4cm) undergone either laparoscopic (n = 112) or open hepatectomy (n = 224) (major hepatectomy accounts for 40.5%), the intraoperative blood loss (median: 159 mL vs. 419 mL), blood transfusion rate (0% vs. 4.5%) and morbidity rate (5.4% vs. 28.1%) were significantly lower in laparoscopic group than open group. The hospital mortality (0% vs. 0.4%), long-term overall (5-year: 56% vs. 42%) and recurrence free (5-year: 36% vs. 33%) survival rates were comparable between groups. (Supplementary information attached) With this experience, the principle investigator proposes an open labelled prospective multi-center randomized trial (AP-LAPO Trial) comparing LMH with OMH for HCC. This study involves 5 high-volume centres specialized in liver surgery and with facilities supporting LMH and OMH in Asia-Pacific region (Hong Kong, Sichuan, Guangzhou and Foshan). These centres perform at least 30 LMH or OMH per year (The Chinese University of Hong Kong, median no. = 51; Kwong Wah Hospital, median no. = 30; West China Medical School of Sichuan University, median no. 120; Eastern Hepatobiliary Surgery Hospital & Institute, median no. = 115; The First People's Hospital of Foshan, median no. = 102), and have achieved excellent perioperative and oncological outcome after LMH or OMH (operative mortality 1% - 2%; complication rate 14% - 23%; 2-year overall survival rate 85% - 88%; 2-year disease-free survival rate 81% - 84%).

Objectives and hypothesis: The primary objective is to test the hypothesis that LMH is associated with less surgical stress, less immunosuppression and thus less tumor recurrence and better survival than OMH. The primary outcome measure is 2-year recurrence-free survival. The secondary outcome measures include hospital mortality, morbidity, quality of life and overall survival between groups. Besides, stress-related cytokines (interleukin-6 [IL-6] and immunosuppressive acidic protein[IAP]) will also be measured during the perioperative

Sample size estimation: Based on a reported 2-year recurrence-free survival rate of 72% after OMH and an expected 88% after LMH (about 20% improvement) according to a previously reported series, 106 patients need to be recruited to each arm in order to demonstrate a statistically significant difference with a 80% power at the 0.05 level of 2-sided significant difference between laparoscopic and open hepatic resection, allowing a drop-out rate of 10%. This sample size will also allow detection of reduction of 2-year tumor recurrence from 50% in OMH group to 30% in LMH with a similar power and level of significance. The principle investigator's unit is a major referral center for management of HCC in Hong Kong, with more than 150 new cases seen per year. There are one other centers in Hong Kong and 3 centers in Mainland China, which are specialized in both laparoscopic and open surgery for patients with HCC, with referral patient number ranging from 50 to 200 per year. The planned number of patients recruited in each participating centres is as follows (The Chinese University of Hong Kong, N = 32; Kwong Wah Hospital, N = 20; West China Medical School of Sichuan University, N = 50; Eastern Hepatobiliary Surgery Hospital & Institute, N = 50; The First People's Hospital of Foshan, median no. = 60) It is therefore expected that recruitment can be completed in about 12 months. All patients will be observed for at least 24 months after treatment. Hence, the total period of study including follow-up is estimated to be about 3 years for the funding period. After the funding period, recruited patients will be followed up periodically up to 5 years after surgery to evaluate the long-term outcome.

Statistical analysis: Statistical analysis will be performed using SPSS version 11.0 (SPSS Inc., Chicago, Ill). The 2-year recurrence-free survival (primary outcome) will be evaluated by Kaplan-Meier method and compared by the log-rank test between studied groups.

Other secondary outcome measures will be compared using Chi-squared test or Fisher's exact test for categorical variables, and Mann-Whitney U test for continuous variables between groups. Overall survival is again computed by the Kaplan-Meier method and compared by the log-rank test between groups. P < 0.05 is considered statistically significant.

Ethical consideration: All aspects of the study will be discussed with each subject during a phone interview or screening visit. An information sheet will be provided, and each subject will be given the opportunity to seek medical advice or to discuss the study with friends or family prior to involvement. Each volunteer will give written, informed consent, in accordance with the attached form, and the subjects will be free to withdraw from the study at any time. This study will be performed in accordance with the ethical standards of the Declaration of Helsinki of 1975 and its later versions. Ethics approval from the institutional review broad of individual center will be sought.

Relevance to clinical applications: The proposed study is an open-labelled prospective multi-center randomized trial investigating the potential benefits of laparoscopic major hepatectomy for hepatocellular carcinoma (HCC), as compared to conventional open surgery. It involves 5 high-volume surgery centers in the Asia-Pacific region, where the incidence of hepatocellular carcinoma is high. The result of this study provides level 1 evidence on the best treatment option for HCC, which needs major hepatectomy. Such information will influence the evidence-based policy in professional practice in the management algorithm for HCC. Since postoperative complications and tumor recurrence are substantial after OMH, potential benefits of LMH tested in this study will help to alleviate these problems. Ultimately, the long-term survival of patients with HCC could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC is in accordance to the diagnostic criteria for HCC used by the European Association for the Study of the Liver. HCC was diagnosed when the radiologic imaging techniques (spiral contrasted CT scan or contrasted MRI) showed typical features of HCC (contrast enhancement in the arterial phase and rapid wash-out of contrast in the venous or delayed phase) and/or elevated serum alpha fetoprotein (AFP) level.
* HCC of maximum diameter up to 10 cm; Single or multiple tumor nodules confined to one liver lobe according to the previous reported series
* Major hepatectomy (resection of > 3 Couinaud's segments) is required as judged by hepatobiliary surgeons
* Absence of extrahepatic metastasis or radiological evidence of venous invasion of major portal vein or hepatic vein branches
* Child's A liver function
* Indocyanine green retention at 15 min (ICG-15) < 15%
* Adequate future liver remnant (image-guided volumetry > 35% of estimated standard liver volume)
* General condition fit for general anaesthesia

Exclusion Criteria:

* Tumors unfavorable for major hepatectomy (e.g. bilobar tumors, main portal vein tumor thrombus and/or inadequate future liver volume)
* Previous treatment for HCC (e.g. transarterial chemoembolization, or chemotherapy)
* Tumors require combined hepatectomy and thermal ablation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival | 2 years
  The proportion of patients surviving without tumor recurrence as measured by postoperative images (CT or MRI) at 2 years

SECONDARY OUTCOMES:
Hospital mortality | 1 year
  Death of patient after index surgery within same hospital admission
Morbidity | 1 year
  Complications of surgery as defined by Clavien-Dindo classification
Quality of llife | 1 year
  Quality of life assessment by Functional Assessment of Cancer Therapy - General questionnaire (Score 0 - 108); high score means good performance status and vice versa
5 - year Overall survival | 5 years
  Overall survival of patients after surgery at 5 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Vogel A, Cervantes A, Chau I, Daniele B, Llovet JM, Meyer T, Nault JC, Neumann U, Ricke J, Sangro B, Schirmacher P, Verslype C, Zech CJ, Arnold D, Martinelli E; ESMO Guidelines Committee. Hepatocellular carcinoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv238-iv255. doi: 10.1093/annonc/mdy308. No abstract available. PMID 30285213
- [Background] Ng KK, Vauthey JN, Pawlik TM, Lauwers GY, Regimbeau JM, Belghiti J, Ikai I, Yamaoka Y, Curley SA, Nagorney DM, Ng IO, Fan ST, Poon RT; International Cooperative Study Group on Hepatocellular Carcinoma. Is hepatic resection for large or multinodular hepatocellular carcinoma justified? Results from a multi-institutional database. Ann Surg Oncol. 2005 May;12(5):364-73. doi: 10.1245/ASO.2005.06.004. Epub 2005 Mar 31. PMID 15915370
- [Background] Hao S, Fan P, Chen S, Tu C, Wan C. Anterior approach to improve the long-term outcome in patients with large-size hepatocellular carcinoma having liver resection. J Surg Oncol. 2016 Dec;114(7):872-878. doi: 10.1002/jso.24433. Epub 2016 Sep 16. PMID 27632953
- [Background] Lee KF, Cheung YS, Wong J, Chong CC, Wong JS, Lai PB. Randomized clinical trial of open hepatectomy with or without intermittent Pringle manoeuvre. Br J Surg. 2012 Sep;99(9):1203-9. doi: 10.1002/bjs.8863. Epub 2012 Jul 24. PMID 22828986
- [Background] Ng KKC, Chok KSH, Chan ACY, Cheung TT, Wong TCL, Fung JYY, Yuen J, Poon RTP, Fan ST, Lo CM. Randomized clinical trial of hepatic resection versus radiofrequency ablation for early-stage hepatocellular carcinoma. Br J Surg. 2017 Dec;104(13):1775-1784. doi: 10.1002/bjs.10677. Epub 2017 Nov 1. PMID 29091283
- [Background] Ng KK, Cheung TT, Pang HH, Wong TC, Dai JW, Ma KW, She WH, Kotewall CN, Lo CM. A simplified prediction model for early intrahepatic recurrence after hepatectomy for patients with unilobar hepatocellular carcinoma without macroscopic vascular invasion: An implication for adjuvant therapy and postoperative surveillance. Surg Oncol. 2019 Sep;30:6-12. doi: 10.1016/j.suronc.2019.05.017. Epub 2019 May 22. PMID 31500787
- [Background] Jarnagin WR, Delman K, Kooby D, Mastorides S, Zager J, Brennan MF, Blumgart LH, Federoff H, Fong Y. Neoadjuvant interleukin-12 immunogene therapy protects against cancer recurrence after liver resection in an animal model. Ann Surg. 2000 May;231(5):762-71. doi: 10.1097/00000658-200005000-00017. PMID 10767798
- [Background] Halls MC, Berardi G, Cipriani F, Barkhatov L, Lainas P, Harris S, D'Hondt M, Rotellar F, Dagher I, Aldrighetti L, Troisi RI, Edwin B, Abu Hilal M. Development and validation of a difficulty score to predict intraoperative complications during laparoscopic liver resection. Br J Surg. 2018 Aug;105(9):1182-1191. doi: 10.1002/bjs.10821. Epub 2018 May 8. PMID 29737513
- [Background] Chen K, Pan Y, Hu GY, Maher H, Zheng XY, Yan JF. Laparoscopic Versus Open Major Hepatectomy for Hepatocellular Carcinoma: A Meta-Analysis. Surg Laparosc Endosc Percutan Tech. 2018 Oct;28(5):267-274. doi: 10.1097/SLE.0000000000000567. PMID 30180140
- [Background] Xu HW, Liu F, Li HY, Wei YG, Li B. Outcomes following laparoscopic versus open major hepatectomy for hepatocellular carcinoma in patients with cirrhosis: a propensity score-matched analysis. Surg Endosc. 2018 Feb;32(2):712-719. doi: 10.1007/s00464-017-5727-2. Epub 2017 Jul 19. PMID 28726140
- [Background] Delvecchio A, Conticchio M, Ratti F, Gelli M, Anelli FM, Laurent A, Vitali GC, Magistri P, Assirati G, Felli E, Wakabayashi T, Pessaux P, Piardi T, Di Benedetto F, de'Angelis N, Briceno-Delgado J, Adam R, Cherqui D, Aldrighetti L, Memeo R. Laparoscopic major hepatectomy for hepatocellular carcinoma in elderly patients: a multicentric propensity score-based analysis. Surg Endosc. 2021 Jul;35(7):3642-3652. doi: 10.1007/s00464-020-07843-7. Epub 2020 Aug 3. PMID 32748269
- [Background] Yoon YI, Kim KH, Kang SH, Kim WJ, Shin MH, Lee SK, Jung DH, Park GC, Ahn CS, Moon DB, Ha TY, Song GW, Hwang S, Lee SG. Pure Laparoscopic Versus Open Right Hepatectomy for Hepatocellular Carcinoma in Patients With Cirrhosis: A Propensity Score Matched Analysis. Ann Surg. 2017 May;265(5):856-863. doi: 10.1097/SLA.0000000000002072. PMID 27849661
- [Background] Marrero JA, Kulik LM, Sirlin CB, Zhu AX, Finn RS, Abecassis MM, Roberts LR, Heimbach JK. Diagnosis, Staging, and Management of Hepatocellular Carcinoma: 2018 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2018 Aug;68(2):723-750. doi: 10.1002/hep.29913. No abstract available. PMID 29624699
- [Background] Abu Hilal M, Aldrighetti L, Dagher I, Edwin B, Troisi RI, Alikhanov R, Aroori S, Belli G, Besselink M, Briceno J, Gayet B, D'Hondt M, Lesurtel M, Menon K, Lodge P, Rotellar F, Santoyo J, Scatton O, Soubrane O, Sutcliffe R, Van Dam R, White S, Halls MC, Cipriani F, Van der Poel M, Ciria R, Barkhatov L, Gomez-Luque Y, Ocana-Garcia S, Cook A, Buell J, Clavien PA, Dervenis C, Fusai G, Geller D, Lang H, Primrose J, Taylor M, Van Gulik T, Wakabayashi G, Asbun H, Cherqui D. The Southampton Consensus Guidelines for Laparoscopic Liver Surgery: From Indication to Implementation. Ann Surg. 2018 Jul;268(1):11-18. doi: 10.1097/SLA.0000000000002524. PMID 29064908
- [Background] Ciria R, Gomez-Luque I, Ocana S, Cipriani F, Halls M, Briceno J, Okuda Y, Troisi R, Rotellar F, Soubrane O, Abu Hilal M. A Systematic Review and Meta-Analysis Comparing the Short- and Long-Term Outcomes for Laparoscopic and Open Liver Resections for Hepatocellular Carcinoma: Updated Results from the European Guidelines Meeting on Laparoscopic Liver Surgery, Southampton, UK, 2017. Ann Surg Oncol. 2019 Jan;26(1):252-263. doi: 10.1245/s10434-018-6926-3. Epub 2018 Nov 2. PMID 30390167
- [Background] Munteanu A, Munteanu D, Iancu M, Lupan I, Samasca G, Aldea C, Mocan T, Iancu C. Assessing immunological surgical stress markers in patients undergoing digestive surgery for pancreatic, hepatic and gastric tumors. J BUON. 2018 Nov-Dec;23(6):1655. PMID 30610790
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] van der Poel MJ, Besselink MG, Cipriani F, Armstrong T, Takhar AS, van Dieren S, Primrose JN, Pearce NW, Abu Hilal M. Outcome and Learning Curve in 159 Consecutive Patients Undergoing Total Laparoscopic Hemihepatectomy. JAMA Surg. 2016 Oct 1;151(10):923-928. doi: 10.1001/jamasurg.2016.1655. PMID 27383568
- [Background] Liu CL, Fan ST, Cheung ST, Lo CM, Ng IO, Wong J. Anterior approach versus conventional approach right hepatic resection for large hepatocellular carcinoma: a prospective randomized controlled study. Ann Surg. 2006 Aug;244(2):194-203. doi: 10.1097/01.sla.0000225095.18754.45. PMID 16858181
- [Background] Ng KKC, Cheng NMY, Huang J, Liao M, Chong CCN, Lee KF, Wong J, Cheung SYS, Lok HT, Fung AKY, Wong GLH, Wong VWS, Lai PBS. Development and validation of a novel nomogram predicting 10-year actual survival after curative hepatectomy for hepatocellular carcinoma. Surgeon. 2021 Dec;19(6):329-337. doi: 10.1016/j.surge.2020.11.013. Epub 2021 Jan 8. PMID 33423927
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Badia JM, Ayton LC, Evans TJ, Carpenter AJ, Nawfal G, Kinderman H, Zografos G, Uemoto S, Cohen J, Habib NA. Systemic cytokine response to hepatic resections under total vascular exclusion. Eur J Surg. 1998 Mar;164(3):185-90. doi: 10.1080/110241598750004625. PMID 9562278
- [Background] Iwanaga T, Suzuki H. Perioperative allogenic blood transfusion and serum levels of immunosuppressive acidic protein in patients undergoing resection of colorectal carcinoma. Dig Dis Sci. 1999 Aug;44(8):1601-4. doi: 10.1023/a:1026619111897. PMID 10492140
- [Background] Igarashi T, Tobe T, Kuramochi H, Akakura K, Ichikawa T, Hamano S, Suzuki N, Furuya Y, Ito H. Serum immunosuppressive acidic protein as a potent prognostic factor for patients with metastatic renal cell carcinoma. Jpn J Clin Oncol. 2001 Jan;31(1):13-7. doi: 10.1093/jjco/hye004. PMID 11256835
- [Background] Shimada M, Takenaka K, Kawahara N, Kajiyama K, Yamamoto K, Shirabe K, Nishizaki T, Yanaga K, Sugimachi K. Surgical treatment strategy for patients with stage IV hepatocellular carcinoma. Surgery. 1996 May;119(5):517-22. doi: 10.1016/s0039-6060(96)80260-1. PMID 8619206
- [Background] Donner A. Approaches to sample size estimation in the design of clinical trials--a review. Stat Med. 1984 Jul-Sep;3(3):199-214. doi: 10.1002/sim.4780030302. PMID 6385187
- [Derived] Ng KKC, Chong CCN, Lee KF, Lai PBS, Cheng TKC, Chen HW, Yi B, Huang JW. Asia-Pacific multicentre randomized trial of laparoscopic versus open major hepatectomy for hepatocellular carcinoma (AP-LAPO trial). BJS Open. 2023 Jan 6;7(1):zrac166. doi: 10.1093/bjsopen/zrac166. PMID 36849753